CLINICAL TRIAL: NCT01978041
Title: Fluoride Bioavailability in Plasma and Saliva After Ingestion of Water or Foods Prepared With Fluoridated Water
Brief Title: Fluoride Bioavailability After Ingestion of Water or Foods Prepared With Fluoridated Water
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Associate Professor, Biochemistry and Cariology, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FOPBioq004
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Dental Caries; Dental Fluorosis
Keywords: pharmacokinetics, saliva, plasma, fluoride, dental fluorosis, dental caries
MeSH Terms: conditions — Dental Caries; Fluorosis, Dental

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Meal prepared with non fluoridated water (<0.1 ppm F) (Experimental)
  Interventions: Other: Meal prepared with non fluoridated water
- Meal prepared with fluoridated water (1 ppm F) (Experimental)
  Interventions: Other: Meal prepared with fluoridated water
- Non fluoridated water (<0.1 ppm F) (Experimental)
  Interventions: Other: Non fluoridated water
- Fluoridated water (1 ppm F) (Experimental)
  Interventions: Other: Fluoridated water
- Pilot study: Meal providing a fluoride dose of 60 ug F/kg (Experimental)
  Interventions: Other: Meal prepared to provide a fluoride dose of 60 ug F/kg
- Pilot study: Meal providing a fluoride dose of 120 ug F/kg (Experimental)
  Interventions: Other: Meal prepared to provide a fluoride dose of 120 ug F/kg

INTERVENTIONS:
Other: Meal prepared with non fluoridated water — Ingestion of a typical brazilian meal (rice, beans, meat, french beans, carrots, gelatin and juice) prepared with purified water containing a fluoride dose of 0.8 ug of fluoride/kg body weight (resulting of the natural fluoride concentration in foods).
  Arms: Meal prepared with non fluoridated water (<0.1 ppm F)
Other: Meal prepared with fluoridated water — Ingestion of a typical brazilian meal (rice, beans, meat, french beans, carrots, gelatin and juice) prepared with fluoridated water (1 ug of fluoride/mL), to provide a total intake of approximately 12 ug of fluoride/kg body weight.
  Arms: Meal prepared with fluoridated water (1 ppm F)
Other: Non fluoridated water — Ingestion of purified water with addition of fluoride to provide a total intake of approximately 0.8 ug of fluoride/kg body weight, which represented the same fluoride ingestion dose of the experimental phase with meal prepared with non fluoridated water.
  Arms: Non fluoridated water (<0.1 ppm F)
Other: Fluoridated water — Ingestion of fluoridated water (1 ug F/mL), to provide a total intake of approximately 12 ug of fluoride/kg body weight.
  Arms: Fluoridated water (1 ppm F)
Other: Meal prepared to provide a fluoride dose of 60 ug F/kg — Ingestion of a typical Brazilian meal (rice, beans, meat, french beans, carrots, gelatin and juice) prepared with non-fluoridated water, with sodium fluoride solution added to the juice to provide a total intake of approximately 60 ug of fluoride/kg body weight.
  Arms: Pilot study: Meal providing a fluoride dose of 60 ug F/kg
Other: Meal prepared to provide a fluoride dose of 120 ug F/kg — Ingestion of a typical Brazilian meal (rice, beans, meat, french beans, carrots, gelatin and juice) prepared with non-fluoridated water, with sodium fluoride solution added to the juice to provide a total intake of approximately 60 ug of fluoride/kg body weight.
  Arms: Pilot study: Meal providing a fluoride dose of 120 ug F/kg

SUMMARY:
The importance of fluoridated water to control caries is well recognized. Although the mode of action of fluoridated water is known (related to a slight increase in fluoride concentration in saliva/dental biofilm in individuals living in fluoridated areas), the kinetics of fluoride concentration in saliva after ingestion of food prepared with fluoridated water, either from fluoride remaining in the oral cavity after mastication, or from fluoride returning from salivary secretion is not known in details. Therefore, the aim of this study is to assess fluoride bioavailability after ingestion of food prepared with fluoridated water. The study will be in vivo, crossover and double blind, in which 12 adult volunteers will participate. In 4 experimental phases, volunteers will ingest: a. a typical Brazilian meal cooked with non-fluoridated water (<0.1 ppm F); b. a typical Brazilian meal cooked with fluoridated water (1 ppm F); c. non fluoridated water (<0.1 ppm F) and d. fluoridated water (1 ppm F). Immediately before and 5, 10, 15, 30, 45, 60, 120, 180 minutes after the ingestion, a blood sample will be collected by digital puncture, and a sample of unstimulated saliva will be collected. Fluoride concentration in the samples will be determined by an ion specific electrode adapted for microanalysis. Results will be analyzed by ANOVA, with significance limit of 5%.

ELIGIBILITY:
Inclusion criteria:

* Good general health
* Good oral health
* Normal salivary flow rate

Exclusion criteria:

* Gastric disorders
* Renal disorders
* Systemic diseases
* Use of drugs that alter salivary flow rate/renal excretion

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma fluoride concentration versus time after water or food ingestion | 180 minutes
  A microsample of blood will be collected by digital puncture before and 5, 10, 15, 30, 45, 60, 120 and 180 min after treatments, to calculate the area under the curve of fluoride concentration in the plasma

SECONDARY OUTCOMES:
Area under the curve of salivary fluoride concentration versus time after water or food ingestion | 180 minutes
  A sample of unstimulated saliva will be collected by digital puncture before and 5, 10, 15, 30, 45, 60, 120 and 180 min after treatments, to calculate the area under the curve of fluoride concentration in saliva
Maximum fluoride concentration in saliva after water or food ingestion | 180 minutes
Maximum fluoride concentration in plasma after water or food ingestion | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Livia MA Tenuta, PhD, Principal Investigator — Piracicaba Dental School, Unversity of Campinas
Locations (1):
- Piracicaba Dental School, University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Falcao A, Tenuta LM, Cury JA. Fluoride gastrointestinal absorption from Na2FPO3/CaCO3- and NaF/SiO2-based toothpastes. Caries Res. 2013;47(3):226-33. doi: 10.1159/000346006. Epub 2012 Dec 29. PMID 23295625
- [Background] Cury JA, Del Fiol FS, Tenuta LM, Rosalen PL. Low-fluoride dentifrice and gastrointestinal fluoride absorption after meals. J Dent Res. 2005 Dec;84(12):1133-7. doi: 10.1177/154405910508401208. PMID 16304442
- [Background] Casarin RC, Fernandes DR, Lima-Arsati YB, Cury JA. [Fluoride concentrations in typical Brazilian foods and in infant foods]. Rev Saude Publica. 2007 Aug;41(4):549-56. doi: 10.1590/s0034-89102006005000034. Portuguese. PMID 17589752